CLINICAL TRIAL: NCT01191086
Title: Open-Label Extension Study to Evaluate the Safety of USL255 as Adjunctive Therapy in Patients With Refractory Partial-Onset Seizures Who Had Participated in P09-004, a Randomized, Multicenter, Double-Blind, Placebo-Controlled, Parallel-Group, Phase 3 Study
Brief Title: Open-label Extension Study to Evaluate the Safety of USL255 in Patients With Refractory Partial-onset Seizures
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Upsher-Smith Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P09-005
Record Dates: First submitted 2010-08-26; First posted 2010-08-30 (Estimated); Results first posted 2015-02-23 (Estimated); Last update posted 2015-02-23 (Estimated); Status verified 2015-02

CONDITIONS: Epilepsy
Keywords: Epilepsy; partial onset seizure; adjunctive therapy
MeSH Terms: conditions — Epilepsy | interventions — Topiramate

ARMS (1):
- Open-label USL255 (Experimental): Topiramate extended-release capsules (USL255) up to a maximum of 400 mg per day
  Interventions: Drug: USL255

INTERVENTIONS:
Drug: USL255
  Other Names: Topiramate extended-release

SUMMARY:
The purpose of this study is to examine the safety of USL255 as adjunctive therapy in patients with refractory partial onset-seizures.

ELIGIBILITY:
Inclusion Criteria:

* Have completed the maintenance period of the P09-004 study.
* Continue to be treated with a stable dose of 1 to a maximum of 3 approved concomitant AEDs.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2010-10; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (68):
- United States (16):
  - Phoenix, Arizona
  - Ventura, California
  - Gainsville, Florida
  - Gulf Breeze, Florida
  - Jacksonville, Florida
  - Port Charlotte, Florida
  - Lexington, Kentucky
  - Waldorf, Maryland
  - Chesterfield, Missouri
  - St Louis, Missouri
  - Somerset, New Jersey
  - Charlotte, North Carolina
  - Toledo, Ohio
  - Dallas, Texas
  - Temple, Texas
  - Milwaukee, Wisconsin
- Argentina (4):
  - Buenos Aires
  - Córdoba
  - Salta
  - Villa Nueva
- Australia (7):
  - Bedford Park
  - Clayton
  - Fitzory
  - Heidelberg West
  - Parkville
  - Randwick
  - Woodville
- Belgium (3):
  - Bruges
  - Duffel
  - Leuven
- Canada (2):
  - Greenfield Park
  - Toronto
- Chile (2):
  - Santiago
  - Valdivia
- Germany (2):
  - Bonn
  - Munich
- Greece (2):
  - Athens
  - Thessaloniki
- India (6):
  - Bangalore
  - Dehradun
  - Hyderabad
  - Mangalore
  - Mumbai
  - New Delhi
- Israel (5):
  - Ashkelon
  - Holon
  - Nahariya
  - Petah Tikva
  - Ramat Gan
- Auckland, New Zealand
- Poland (6):
  - Gdansk
  - Katowice
  - Krakow
  - Lodz
  - Lublin
  - Warsaw
- Russia (6):
  - Kazan'
  - Moscow
  - Saint Petersburg
  - Samara
  - Tyumen
  - Yaroslavi
- Cape Town, South Africa
- Spain (5):
  - Badalona
  - Barakaldo
  - Granada
  - Madrid
  - Valencia

REFERENCES:
- [Derived] Chung SS, Hogan RE, Blatt I, Lawson P B, Nguyen H, Clark AM, Anders B, Halvorsen MB; PREVAIL OLE Study Group. Long-term safety and sustained efficacy of USL255 (topiramate extended-release capsules) in patients with refractory partial-onset seizures. Epilepsy Behav. 2016 Jun;59:13-20. doi: 10.1016/j.yebeh.2016.03.005. Epub 2016 Apr 14. PMID 27084978

RESULTS

PARTICIPANT FLOW:
Groups:
- Open-label USL255: Topiramate extended-release capsules (USL255) up to a maximum of 400 mg per day
  USL255
Period: Overall Study
Arm/Group | Open-label USL255
Started | 210
Completed | 148
Not Completed | 62
Not completed — Adverse Event | 20
Not completed — Lack of Efficacy | 10
Not completed — Lost to Follow-up | 4
Not completed — Physician Decision | 2
Not completed — Withdrawal by Subject | 24
Not completed — Discontinuation criterion met | 1
Not completed — Other | 1

BASELINE CHARACTERISTICS:
Arm/Group | Open-label USL255
Number analyzed (Participants) | 210
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.5 (11.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 114
  Male | 96

OUTCOME MEASURES:

1. Primary Outcome: Evaluate the Safety of USL255 Through the Collection of Adverse Events and Clinical Laboratory Evaluations
Time Frame: Open label treatment of up to 62 weeks
Population: The intent-to-treat (ITT) population was used for all analyses. The ITT population included all subjects who received at least 1 dose of study drug in this extension study.
Measure: Number; unit: participants
Arm/Group | Open-label USL255
Number analyzed (Participants) | 210
participants
  No. of participants analyzed | 210
  No. with ≥ 1 treatment-emergent AE | 146
  No. with ≥ 1 treatment-related AE | 102
  No. with severe AEs | 15
  No. with serious AEs | 14
  No. with TEAEs leading to study discontinuation | 20
  No. of deaths related to study drug | 0
  No. of deaths unrelated to study drug | 1

ADVERSE EVENTS:
Time Frame: Open-label treatment of up to 62 weeks
Description: Safety of adjunctive USL255 was assessed through collection of adverse events (AEs) reports and clinical laboratory evaluations during the open-label treatment study
Arm/Group | Open-label USL255
Serious Adverse Events (participants affected / at risk) | 14/210
Other Adverse Events (participants affected / at risk) | 61/210
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Open-label USL255 (N=210)
Cholelithiasis (Hepatobiliary disorders) | 2
Cholecystitis acute (Hepatobiliary disorders) | 1
Status epilepticus (Nervous system disorders) | 2
Convulsion (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Ischaemic stroke (Nervous system disorders) | 1
Acute psychosis (Psychiatric disorders) | 1
Appendicitis (Infections and infestations) | 1
Diarrhea infectious (Infections and infestations) | 1
Lobar pneumonia (Infections and infestations) | 1
Balance disorder (General disorders) | 1
Fibula fracture (Injury, poisoning and procedural complications) | 1
Tibia fracture (Injury, poisoning and procedural complications) | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1
Volvulus (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Open-label USL255 (N=210)
Somnolence (Nervous system disorders) | 15
Dizziness (Nervous system disorders) | 13
Aphasia (Nervous system disorders) | 11
Weight decreased (Investigations) | 16
Headache (Nervous system disorders) | 16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No